CLINICAL TRIAL: NCT06794580
Title: The Interplay Between Emotional Processing and Self-Monitoring in Neurodegenerative Patients
Brief Title: The DUAL-SYSTEM HYPOTHESIS of ANOSOGNOSIA: the Interplay Between Emotional Processing and Self-Monitoring in Neurodegenerative Patients
Acronym: ASSESS
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C17-77
Record Dates: First submitted 2019-01-17; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anosognosia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Controls: One group of 40 cognitively healthy controls (MMSE score, >27; CDR score, 0; education-, gender-, and aged-matched) that will be recruited among patients' spouses and from the community.
- Frontotemporal Dementia: One group of 30 patients fulfilling the core diagnostic features of bvFTD;
- ALZHEIMER DISEASE: One group of 30 patients fulfilling the core diagnostic features of AD.

SUMMARY:
The ASSESS project is a monocenter, regionally based, study evaluating the pathophysiological/functional processes underlying anosognosia in both AD and bvFTD. The multimodal analysis will be applied to the obtained cognitive, neuroimaging and electrophysiological data in order to describe the mechanistic cascade of anosognosia and their neuronal and electrophysiological biomarkers. Importantly, it has the potential to significantly impact society by: i) addressing a fundamental scientific question towards a causal understanding on how self-awareness emerges in the human brain; and ii) developing a cognitive BCI-system, which will allow us to validated neurophenomenologically EEG biomarkers in anosognosia, and may give us access in later steps to neurofeedback applications for the improvement of self-awareness in early stages of AD and bvFTD, with major social and economic gains.

DETAILED DESCRIPTION:
1. INTRODUCTION The ability to appraise our own performance is a unique component of human functioning. It is impaired in brain diseases responsible for anosognosia, resulting in poor self-appraisal of one's own deficits. Anosognosia negatively impacts on capacity issues, such as treatment compliance and the patients' ability to deal appropriately with risk situations, with damaging consequences on their quality of life. Furthermore, it places a serious burden on the healthcare systems and may be extremely distressing for the patients' caregivers. Although initially described after vascular brain lesions and frequently observed in neurodegenerative disorders, such as the Alzheimer's disease (AD) or the behavioral variant of frontotemporal dementia (bvFTD), anosognosia remains an intriguing phenomenon and its neural mechanisms largely unknown. There is, however, evidence in neurodegenerative disorders pointing to frontally-mediated dysfunctions as causes of anosognosia. Here, we build on a convergence of emotional and self-monitoring processes, and specifically explore their role in the emergence of anosognosia in AD and bvFTD patients, thus predicting that unawareness across domains may depend on common processes. In particular, we hypothetize that anosognosia might result from the inability to establish the linkage between emotional arousal and self-monitoring (that would normally trigger adaptive behaviors), due to critical connectivity impairments in the uncinate fasciculus in both AD and bvFTD (regardless to the nature of the deficits to which the patients are unaware). Indeed, by virtue of its connectivity, linking limbic with frontal/executive systems, one might expect that the uncinate fasciculus plays a major role in the interplay between emotional arousal and self-monitoring.
2. OBJECTIVES

The main scientific, clinical and technological objectives of this project are:

1. To test the interplay between self-monitoring and autonomic reactivity (as a proxy of emotional arousal) and then determine whether it is disturbed in both groups of patients relative to healthy controls, and whether it correlates with the patients' anosognosia level, as measured by standard scales (STUDY 1);
2. To test whether structural and functional damage to the uncinate fasciculus correlate with the patients' anosognosia level, and whether it may be critical for the emergence of this neurological syndrome (STUDY 2); and
3. To establish the neurophysiological markers of anosognosia in order to further develop a cognitive Brain-computer interface (BCI) aimed at monitoring patients' self-awareness in real time (STUDY 3).

3. PROJECT IMPLEMENTATION

The current project will be implemented over three distinct periods, corresponding to 3 well-identified work packages (WPs), during 48 months: 1. Data Acquisition; 2. Data Analysis; and 3. BCI Application WPs, as follows:

1. Data Acquisition: This WP 1 corresponds to a 24-months period that will be devoted to participants' recruitment, including both patients and healthy controls; and data acquisition, including behavioral, electrophysiological and neuroimaging data. Behavioral and electrophysiological data will be collected at the IM2A, whereas neuroimaging data will be acquired at the center for neuroimaging research (CENIR), both at the Salpêtrière's hospital, in Paris.
2. Data Analysis: This WP 2 corresponds to an 18-months period (partially overlapping with the WP1), during which we will be aimed at analyzing the acquired new data and further developing the functional and mechanistic foundations of the findings, as well as their theoretical and practical implications. During this period, we will also work on the discussion and publication of preliminary findings.
3. BCI Application: This WP 3 corresponds to the last 12-months period of the project; the main focus will be on the development of a cognitive BCI-system specifically targeting anosognosia. In parallel, we will continue working on the publication and dissemination of the project results.
4. METHODS Participants An hundred (n=100) native French speakers, age 50 years or above, with normal color vision and with normal or corrected-to-normal visual acuity, will be recruited for the project. A signed informed consent will be obtained from all participants, as well as from the patients' caregivers.

   Patients : Two groups of patients (n=60) will be recruited at the Institut de la Mémoire et de la Maladie d'Alzheimer of the Salpêtrière's hospital, as follows: 1. One group of 30 patients fulfilling the core diagnostic features of bvFTD (Rascovsky et al, 2011); and 2. One group of 30 patients fulfilling the core diagnostic features of AD (Dubois et al, 2014), both in a mild cognitive and functional severity stage, as determined by a Mini-Mental Status Examination (MMSE; Folstein et al, 1975) score greater than or equal to 18, and a Clinical Dementia Rating scale (CDR; Hughes et al, 1982; Morris, 1993) global score less than or equal to 2.

   The other group corresponds to 40 cognitively healthy controls (MMSE score, >27; CDR score, 0; education-, gender-, and aged-matched) that will be recruited among patients' spouses and from the community.

   Neuropsychological tests In addition to the MMSE and the CDR, patients will be administered the frontal assessment battery (FAB; Dubois et al, 2000), as well as neuropsychological tests of verbal episodic memory (Grober & Buschke, 1987), short term memory (digit span), phonemic and semantic verbal fluency, visual-spatial function and calculations. Patients' mood will be assessed with both the Hamilton Rating Scale for Depression (Hamilton, 1960) and the Geriatric Depression Scale (Yesavage et al, 1983; Greenberg, 2007), while apathy will be assessed with the Neuropsychiatric Inventory (NPI; Cummings et al, 1994).

   Anosognosia measures Patients level of self-appraisal accuracy will be evaluated by using i) patient-informant questionnaires designed to assess both episodic memory and executive functions' abilities, as well as activities of daily living (Migliorelli et al,1995; Dalla Barba et al, 2015); and ii) patients' postdiction-performance (Fragkiadaki et al, 2016) approaches.

   Neuroimaging and electrophysiological techniques An EEG and a brain MRI will also be administered to the patients (AD and bvFTD) and the healthy controls. In particular, our methodological approach will combine behavioral with advanced electrophysiological and neuroimaging methods that all tap on self-monitoring abilities and their relation to both emotional arousal and measures of self-appraisal accuracy. Importantly, recent evidence supports the brain's ability to modify and learn even in early stages of dementia, which may thus constitute a critical window for Brain Computer-Interfaces (BCI) interventions in neurodegenerative patients. Typically, BCIs acquire brain waves from an EEG amplifier and then utilize the biomarkers derived from the brain signal and adapt to the user's performance. The goal is to apply neuro-physiological regulation to foster cortical reorganization, thus promoting neural plasticity. The development of a cognitive BCI monitoring anosognosia is a necessary step to design specific neurofeedback strategies improving self-awareness, even though considerable development and controlled clinical trials will be required before these BCI interventions earn a place in our standard of clinical care.

   Exclusion criteria for all participants are: i) prior neurological disease or neurosurgery; ii) report of a present or prior major psychiatric disorder; iii) potentially confounding medications, particularly those with effects on the peripheral nervous system; and iv) contraindication for magnetic resonance imaging.
5. OPERATIONAL PART OF THE PROTOCOL Cognitive and electrophysiological data will be collected at the Institut de la Mémoire et de la Maladie d'Alzheimer (IM2A) during the first visit (V1), whereas neuroimaging data will be acquired at the Center for Neuroimaging Research (CENIR) during the second and last visit (V2), both at the Salpêtrière's hospital, in Paris. The V2 must take place 1 day up to 3 months after the V1.

First visit (V1): The V1 is also the screening visit and all assessments to be performed at this visit are shown in the study flow-chart, section 3. Both the cognitive/behavioural and EEG data will be acquired at the IM2A. The complete visit will last approximately 3h30min.

Second visit (V2): The V2 will take place one day up to three months after the V1.

During this visit, both patients and controls will be administered a brain MRI (structural and functional). This MRI will be performed using a 3 Tesla Scanner at the CENIR, in the Salpêtrière's hospital. A custom-built head holder will be used to prevent head movement. Both resting-state BOLD images and DTI images will be acquired using SENSE acquisition, 45 min total imaging time.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS and HEALTHY CONTROLS :

* French speakers*, age ≥ 50 ≤ 85 years of age, with normal color vision or corrected-tonormal visual acuity,
* Capacity to consent,
* Covered by social security,
* Ability to undergo MRI scanning,
* The spouse / caregiver is able to accompany the subject to both visits and ready to complete questionnaires.
* Already in menopause (for women)

PATIENTS :

30 patients fulfilling the core diagnostic features of bvFTD; 30 patients fulfilling the core diagnostic features of AD; both in a mild to moderate cognitive and functional severity stage, as determined by: MMSE score greater than or equal to 18, and CDR global score less than or equal to 2, Grober et Buschke: TRGB < 42 as well as clinical signs (subjective impression) of anosognosia.

HEALTHY SUBJECTS (n=40) :

MMSE score ≥ 27;TRGB> 42 Education, gender-, and aged-matched controls. * Subjects will be administered neuropsychological tests that have been validated for French speakers.

Exclusion Criteria:

* Illiteracy /unable to count or to read;
* Having a neurological disorder, such as: epilepsy, extrapyramidal signs, brain tumour, subdural haematoma, history of head trauma followed by persistent neurological deficits (motor, sensory or cognitive); stroke that has occurred in the last three months;
* Report of a present or prior major psychiatric disorder;
* Potentially confounding medications, particularly beta-blockers that may have effects on the peripheral nervous system; typically, beta-blockers are used to control heart rhythm, treat angina, and reduce high blood pressure.
* Person deprived of their liberty by judicial or administrative decision
* Participation in a drug trial or exclusion period of another study
* Inability to understand information about the protocol
* Meeting brain MRI exclusion criteria (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body, claustrophobia) or refusing MRI. * Contra-indication questionnaire to be filled in beforehand.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to recruit a total of 100 subjects, including 30 patients with bvFTD, 30 patients with AD, and 40 healthy, age-, gender-, and education level-matched controls.
  Since the project aims at investigating the mechanistic cascade that makes bvFTD and AD patients to become unaware of their deficits, the testing of such patients and healthy controls is necessary.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
ELECTROPHYSIOLOGICAL AND ELECTRODERMAL MEASURES | 45 Minutes
  Primary studied parameters include the measure of:
  i) A classic marker of brain responses to one's own errors, which can be measured by EEG (the so-called error-related negativity, ERN), regarding the individual variability and between-group differences in self-monitoring accuracy;
  ii) The ERN amplitude and latency, as indexes of self-monitoring ability, regarding subjects' emotional arousal, as studied by the amplitude of electrodermal responses (EDRs);
  iii) The ERN amplitude and latency, and the EDR amplitudes, regarding the level of anosognosia within the patients' groups.

SECONDARY OUTCOMES:
NEUROIMAGING | 45 minutes
  Secondary studied parameters include:
  i) Between-group analysis of subjects' measures of the uncinate fasciculus integrity;
  ii) Measures of the uncinate fasciculus integrity regarding individual scores on anosognosia tests and other measures of self-monitoring tasks among the patients' groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de la Mémoire et de la Maladie d'Alzheimer (IM2A), Paris, paris, France

IPD SHARING:
Plan to Share IPD: No